CLINICAL TRIAL: NCT01039623
Title: Randomized Assessment of Safety and Immunogenicity of Intradermal Unadjuvanted Portion of Pandemrix® Via a Microneedle Device With Intramuscular Adjuvanted Pandemrix® as Reference
Brief Title: Assessment of Safety and Immunogenicity of Intradermal Unadjuvanted Portion of Pandemrix® Via a Microneedle Device With Intramuscular Adjuvanted Pandemrix® as Reference
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Engelhard Dan, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vaccine-HMO-CTIL
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2009-12

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — pandemrix

INTERVENTIONS:
Biological: Pandemrix® (H1N1 pandemic influenza) — vaccinated against H1N1 pandemic influenza. One group will receive the adjuvant vaccine while the other group will get intradermal antigen, without the adjuvant.

SUMMARY:
Healthy volunteers will be vaccinated against H1N1 pandemic influenza. One group will receive the adjuvant vaccine while the other group will get intradermal antigen, without the adjuvant. The antibody production will be compared.

DETAILED DESCRIPTION:
Healthy volunteers will be vaccinated against H1N1 pandemic influenza. One group will receive the adjuvant vaccine while the other group will get intradermal antigen, without the adjuvant. The antibody production will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-64
* Both genders
* Healthy

Exclusion Criteria:

* Under 18 or above 64
* Not healthy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
antibody levels | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel